CLINICAL TRIAL: NCT02352337
Title: Randomised Phase II Study in Metastatic Pancreatic Cancer Evaluating FOLFIRINOX +/- LV5FU2 in Maintenance Versus Firgem in First-line
Brief Title: First-line Metastatic Pancreatic Cancer : FOLFIRINOX +/- LV5FU2 in Maintenance Versus Firgem
Acronym: PANOPTIMOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE35
Record Dates: First submitted 2015-01-14; First posted 2015-02-02 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: cancer; pancreatic cancer; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — folfirinox; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FOLFIRINOX (Active Comparator): Every two weeks (maximum of 12 cycles) : Oxaliplatin 85 mg / m2 Day1 in 2 hours - then Irinotecan 180 mg / m2 Day1 in 90 minutes - Folinic acid 400 mg / m2 Day1 in 2 h (during the irinotecan infusion) - 5-FU bolus 400 mg / m² Day1 followed by continuous 5-FU 2400 mg / m2 total over 46 hours
  Interventions: Drug: FOLFIRINOX
- FOLFIRINOX + LV5FU2 in maintenance (Experimental): Folfirinox during 4 months followed by LV5FU2 maintenance until progression:
  Folfirinox (as described in arm FOLFIRINOX) LV5FU2 : Folinic acid 400 mg/m² (200 mg/m² if Elvorine), in perfusion over 2 hours the 5FU 400 mg/m² in bolus over 10 mn followed by 5FU 2400 mg/m² in perfusion over 46 hours.
  Interventions: Drug: FOLFIRINOX; Drug: LV5FU2
- FIRGEM (Experimental): Alternance of 2 months of FOLFIRI.3 with 2 months of GEMCITABINE:
  Folfiri.3: Irinotécan 90 mg/m² at day 1 in perfusion over 60 minutes in parralel of folinic acid Folinic acid 400 mg/m² (or 200 mg/m² Elvorine) at day 1 in perfusion over 2 hours 5FU continue 2000 mg/m² over 46 heures then irinotécan at 90 mg/m² (1h) at day 3 when 5U perfusion is over
  Gemcitabine: 1000 mg/m² in perfusion over 30 mn at day 1,8,15,29,36 and 43 over (1 injection per week during 3 weeks followed with 7 days of rest )
  Interventions: Drug: FOLFIRI.3; Drug: Gemcitabine

INTERVENTIONS:
Drug: FOLFIRINOX — Perfusion :oxaliplatine, Irinotecan ,folinic acid, 5FU bolus and continue
  Arms: FOLFIRINOX; FOLFIRINOX + LV5FU2 in maintenance
Drug: LV5FU2 — Perfusion: Folinic Acid,5FU Bolus,5FU continue
  Arms: FOLFIRINOX + LV5FU2 in maintenance
Drug: FOLFIRI.3 — Perfusion :Irinotecan,Acide folinique ,5FU continue
  Arms: FIRGEM
Drug: Gemcitabine — Gemcitabine perfusion
  Arms: FIRGEM

SUMMARY:
The pancreas cancer is the 4th cause of death. All stage confused, the survival at 5 years is note over 5 %. At metastatic stage, the pancreatic adenocarcinoma is an incurable disease with the survival median of 2-4 months without chemotherapy.

Up to 2011, gemcitabine was the only reference treatment of this type of cancer. But until, the FOLFIRINOX could permitted to improve significantly the overall survival (6,8 months with gemcitabine vs 11,1 months with FOLFIRINOX) and the progression free survival (3,3 months with gemcitabine vs 6,4 months with FOLFIRINOX) for patients under 76 years. Main toxicities of this treatment are hematological, gastrointestinal and neuropathy with apparition of sensitive neuropathy, reversible, related to oxaliplatin.

These results are on a population under 76 years old. In this study, the median age of patients at inclusion was 61 years old and FOLFIRINOX was still beneficial for patients more than 65 years old. Given the increase of proportion of patients than more of 65 years old with pancreatic cancer and given the increase of life expected, it is important to know the effectiveness and tolerance of such treatment for patient older than 65 years and 76 years.

FIRGEM is an original strategic sequential treatment witch alternates, every 2 month, 4 cycles of FOLFIRI.3 and 2 cycles of 3 injections of gemcitabine. There is no cross resistance known between this 2 treatments witch limit toxicities and preserve quality of life of patients. A Phase II trial testing this treatment regimen to classical regimen of gemecitabine, showed an overall survival of 11 months in the FIRGEM regimen and an overall survival of 8,2 months in the gemcitabine regimen. The rate of progression was 45% near of progression rate with FOLFIRINOX. Tolerance is close to that FOLFIRINOX regimen but this strategic doesn't induce limiting neurotoxicities and allow to use oxaliplatin in 2de line of treatment.

The trial propose to evaluate the effectiveness and tolerance of FOLFIRINOX regimen (8 cycles) with LV5FU2 in maintenance (that could increase the FOLFIRINOX tolerable without decrease efficiency), to FIRGEM regimen and to FOLFIRINOX (12 cycles) which is the reference regimen.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease
* At least one mesurable lesion according to RECIST V1.1 criteria
* No prior chemotherapy (excepted if there is at least on lestion out of the irradition area)
* Age > 18 years. A favorable adviced by an onco geriatrician would be mandatory for inclusion of patients older than 75 older
* Performance statut (WHO) 0-1
* Polynyclear ≥ 1500/mm3
* Bilirubine ≤ 1,5 fois la LSN, creatinin < 120μmol / L
* Signed informed consent form

Exclusion Criteria:

* Another type of pancreas tumor, as endocrine tumor ou with acinous cells
* Ampulloma
* Cerebral or meningeal metastasis
* Gilbert disease
* Neuropathie > or = grade 1
* Study treatments contraindication
* Uncontrolled diarrhoea or inflamatory disease of colon or rectum, or bowel obstruction or bowel sub-obstruction no resolved with specific treatment
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease prevent patient to receive study Cancer within the 5 years before inclusion, except for int situ cancer of the neck of the uterus or basal cell skin cancer
* Significant previous cardiac and respiratory disease
* Patient included in an other therapeutic study with experimental treatment
* Pregnancy or breast feeding
* Patient depreved of freedom or under gardianship
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DAHAN Laetitia, MD, Principal Investigator — MARSEILLE La Timone
Locations (54):
- France (54):
  - CHU - Hôtel Dieu, Angers
  - CH, Auxerre
  - CH - Henri Duffaut, Avignon
  - Centre d'oncologie et de radiothérapie, Bayonne
  - CH, Bayonne
  - Ch - Ch Beauvais, Beauvais
  - CHU, Besançon
  - Bezier Ch, Béziers
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord, Bordeaux
  - CH -Duchenne, Boulogne-sur-Mer
  - CHU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - CH Compiègne-Noyon, Compiègne
  - CHG, Corbeil-Essonnes
  - CHU - Hôpital François Mitterand, Dijon
  - CH, Dunkirk
  - CHU de Grenoble, Grenoble
  - Institut Daniel Hollard / Groupe Hospitalier Mutualiste, Grenoble
  - Clinique Sainte Marguerite, Hyères
  - CH Marne La Vallée Jossigny, Jossigny
  - CHD, La Roche-sur-Yon
  - CHU - Claude Huriez, Lille
  - Hôpital du Scorff, Lorient
  - CHU - Hôpital Edouard Herriot, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - La Timone, Marseille
  - Hôpital Européen de Marseille, Marseille
  - Hôpital privé, Marseille
  - CH - Centre Hospitalier de Meaux, Meaux
  - Centre Antoine Lassagne, Nice
  - Hôpital de la Source -service HGE et cancérologie digestive, Orléans
  - Hôpital de la Source- service d'oncologie, Orléans
  - CHU AP - HP - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Saint Joseph, Paris
  - Hôpital La Pitié Salpetière, Paris
  - CH Pau, Pau
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHU Robert Debré, Reims
  - Centre Eugène Marquis, Rennes
  - CHU - Charles Nicolle, Rouen
  - CHU, Saint-Etienne
  - CH, Soissons
  - CH, St-Malo
  - Centre Paul Strauss, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - CH - Bigorra, Tarbes
  - Hôpityal Trousseau, Tours
  - CH, Valenciennes
  - Institut Gustave Roussy, Villejuif
  - Hôpital Privé de Villeneuve d'Ascq, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dahan L, Williet N, Le Malicot K, Phelip JM, Desrame J, Bouche O, Petorin C, Malka D, Rebischung C, Aparicio T, Lecaille C, Rinaldi Y, Turpin A, Bignon AL, Bachet JB, Seitz JF, Lepage C, Francois E; PRODIGE 35 Investigators/Collaborators. Randomized Phase II Trial Evaluating Two Sequential Treatments in First Line of Metastatic Pancreatic Cancer: Results of the PANOPTIMOX-PRODIGE 35 Trial. J Clin Oncol. 2021 Oct 10;39(29):3242-3250. doi: 10.1200/JCO.20.03329. Epub 2021 Jul 21. PMID 34288696
- [Derived] Boisteau E, Dahan L, Williet N, Le Malicot K, Desrame J, Bouche O, Petorin C, Malka D, Rebischung C, Aparicio T, Lecaille C, Rinaldi Y, Turpin A, Bignon AL, Bachet JB, Lepage C, Granger V, Legoux JL, Deplanque G, Baconnier M, Lecomte T, Bonnet I, Seitz JF, Francois E, Lievre A; PRODIGE 35 Investigator/Collaborators. Clinico-biological factors predicting the benefit of the LV5FU2 maintenance strategy as a first-line therapy in patients with metastatic pancreatic cancer. Oncologist. 2024 Sep 6;29(9):e1149-e1158. doi: 10.1093/oncolo/oyae079. PMID 39235326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 276 patients were randomized by 53 centers in France between 12 January 2015 and 28 November 2016.
  3 patients withdrew their consent so they were never part on analyses populations.
Groups:
- FOLFIRINOX + LV5FU2 in Maintenance: Folfirinox during 4 months followed by LV5FU2 maintenance until progression:
  Folfirinox (as described in arm FOLFIRINOX) LV5FU2 : Folinic acid 400 mg/m² (200 mg/m² if Elvorine), in perfusion over 2 hours the 5FU 400 mg/m² in bolus over 10 mn followed by 5FU 2400 mg/m² in perfusion over 46 hours.
  FOLFIRINOX: Perfusion :oxaliplatine, Irinotecan ,folinic acid, 5FU bolus and continue
  LV5FU2: Perfusion: Folinic Acid,5FU Bolus,5FU continue
- FIRGEM: Alternance of 2 months of FOLFIRI.3 with 2 months of GEMCITABINE:
  Folfiri.3: Irinotécan 90 mg/m² at day 1 in perfusion over 60 minutes in parralel of folinic acid Folinic acid 400 mg/m² (or 200 mg/m² Elvorine) at day 1 in perfusion over 2 hours 5FU continue 2000 mg/m² over 46 heures then irinotécan at 90 mg/m² (1h) at day 3 when 5U perfusion is over
  Gemcitabine: 1000 mg/m² in perfusion over 30 mn at day 1,8,15,29,36 and 43 over (1 injection per week during 3 weeks followed with 7 days of rest )
  FOLFIRI.3: Perfusion :Irinotecan,Acide folinique ,5FU continue
  Gemcitabine: Gemcitabine perfusion
Period: Overall Study
Arm/Group | FOLFIRINOX | FOLFIRINOX + LV5FU2 in Maintenance | FIRGEM
Started | 91 | 92 | 90
Completed | 87 | 91 | 88
Not Completed | 4 | 1 | 2
Not completed — Patients never treated | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented on the ITT population meaning all the randomized patients who have not withedrew their consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFIRINOX | FOLFIRINOX + LV5FU2 in Maintenance | FIRGEM | Total
Number analyzed (Participants) | 91 | 92 | 90 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 51 | 41 | 138
  >=65 years | 45 | 41 | 49 | 135
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.55 [55.78 to 69.53] | 64.18 [59.61 to 68.77] | 65.88 [59.73 to 70.26] | 64.81 [59.08 to 69.54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 43 | 112
  Male | 56 | 58 | 47 | 161
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 91 | 92 | 90 | 273
Region of Enrollment [Number; unit: participants]
  France | 91 | 92 | 90 | 273

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive and Without Radiological and/or Clinical Progression 6 Months After the Randomization.
Description: Progression was defined as radiological progression according to RECIST v1.1 criteria and/or clinical progression according to the investigator. Progression or death (for any reason) was considered if the event occured within the first 6 months since randomization. 6 month scans were 6 month scans with a +/- 1 month window.
Time Frame: 6 months after randomization
Population: The primary endpoint was analysed on the mITT population meaning all the randomized patients with at least one dose of study drug taken
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX | FOLFIRINOX + LV5FU2 in Maintenance | FIRGEM
Number analyzed (Participants) | 87 | 91 | 88
Participants | 41 | 39 | 30

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the patient's death (all causes). For alive patients, the date of last news was taken into account.
  The analysis was done on the ITT population meaning the patients who have been randomized. Numbers of patients correspond the number of patients randomized in the study.
Time Frame: Up to 3 years after the treatment start
Population: Endpoint was analyzed on the ITT population meaning the patients randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRINOX | FOLFIRINOX + LV5FU2 in Maintenance | FIRGEM
Number analyzed (Participants) | 91 | 92 | 90
months | 10.09 [8.54 to 12.16] | 11.20 [9.03 to 13.14] | 7.34 [5.72 to 9.49]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: It was defined as the time between t randomization and the date of the first radiological progression (RECIST 1.1 criteria) and/or clinical progression according to the investigator or death (whatever the cause is); Patients alive without progression were censored at date of last news
  .
Time Frame: up to 12 months after randomization
Population: The analysis was done on the ITT population meaning the patients who have been randomized into the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRINOX | FOLFIRINOX + LV5FU2 in Maintenance | FIRGEM
Number analyzed (Participants) | 91 | 92 | 90
months | 6.28 [5.32 to 7.56] | 5.73 [5.26 to 7.29] | 4.50 [3.48 to 5.72]

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 3 years but adverse Events were assessed up to 1 year.
Description: Adverse events were analyzed on the population of patients who received at leats one dose of treatment and regarding the treatment really received by the patient. One patient randomized in the FIRGEM arm recieved FOLFIRINOX. So, this patient was analyzed in the Folfirinox arm for tolerance
  For all cause of mortality, the population was the ITT population meaning all patients randomized.
Arm/Group | FOLFIRINOX | FOLFIRINOX + LV5FU2 in Maintenance | FIRGEM
All-Cause Mortality (participants affected / at risk) | 82/91 | 80/92 | 83/90
Serious Adverse Events (participants affected / at risk) | 31/88 | 53/91 | 57/87
Other Adverse Events (participants affected / at risk) | 88/88 | 91/91 | 87/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRINOX (N=88) | FOLFIRINOX + LV5FU2 in Maintenance (N=91) | FIRGEM (N=87)
Diarrhea (Gastrointestinal disorders) | 6 | 8 | 8
Abdominal pain (Gastrointestinal disorders) | 3 | 10 | 11
Vomiting (Gastrointestinal disorders) | 9 | 8 | 9
Naus (Gastrointestinal disorders) | 2 | 3 | 5
Catheter infection (Infections and infestations) | 1 | 3 | 2
Septicemia (Infections and infestations) | 2 | 5 | 8
Anemia (Investigations) | 3 | 1 | 2
PNN decrease (Investigations) | 1 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 7
Fatigue (General disorders) | 8 | 16 | 15
Fever (General disorders) | 3 | 4 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRINOX (N=88) | FOLFIRINOX + LV5FU2 in Maintenance (N=91) | FIRGEM (N=87)
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 21 | 20
Palmo-plantar syndrome (Skin and subcutaneous tissue disorders) | 5 | 18 | 3
Dysgueusia (Nervous system disorders) | 3 | 9 | 3
Neurotoxicity (Nervous system disorders) | 68 | 70 | 8
Constipation (Gastrointestinal disorders) | 28 | 31 | 28
Diarrhea (Gastrointestinal disorders) | 66 | 71 | 67
Abdominal pain (Gastrointestinal disorders) | 33 | 41 | 42
Mucitis (Gastrointestinal disorders) | 31 | 30 | 18
Nausea (Gastrointestinal disorders) | 65 | 74 | 64
Vomiting (Gastrointestinal disorders) | 42 | 50 | 52
Dorsalgia (Musculoskeletal and connective tissue disorders) | 6 | 12 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 3
Anorexia (Metabolism and nutrition disorders) | 42 | 54 | 50
Fatigue (General disorders) | 74 | 78 | 74
Fever (General disorders) | 12 | 29 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-08-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02352337/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT02352337/SAP_001.pdf